CLINICAL TRIAL: NCT00843973
Title: Osteogenic Cell Viability in Bone Graft Obtained Using the Reamer Irrigator Aspirator (RIA) System Versus Iliac Crest Bone Graft
Brief Title: Osteogenic Cell Viability in Bone Graft
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: AO North America (Other)
Responsible Party: Principal Investigator, Brett Crist, Assistant Professor, Co-Director of Trauma Services, Co-Director Orthopaedic Trauma Fellowship, Department of Orthopaedic Surgery, University of Missouri-Columbia
Other Study IDs: IRB 1095798
Record Dates: First submitted 2009-01-26; First posted 2009-02-13 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Fractures, Closed
Keywords: Iliac Crest Bone Graft; Reamer Irrigator Aspirator
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- iliac crest bone graft: Bone graft harvested via iliac crest bone graft procedure
  Interventions: Procedure: iliac crest bone graft
- Reamer Irrigator Aspirator: Bone graft harvested via the Reamer Irrigator Aspirator (RIA) Procedure
  Interventions: Procedure: Reamer Irrigator Aspirator

INTERVENTIONS:
Procedure: iliac crest bone graft — iliac crest bone graft procedure
  Other Names: ICBG
  Groups: iliac crest bone graft
Procedure: Reamer Irrigator Aspirator — Reamer Irrigator Aspirator (RIA) Procedure
  Other Names: RIA
  Groups: Reamer Irrigator Aspirator

SUMMARY:
The purpose of this study is to find out if the cells in bone graft samples collected using a reamer are similar to the cells in bone graft samples collected using the iliac crest bone graft method.

DETAILED DESCRIPTION:
Although iliac crest bone grafting is the gold standard for autogenous bone grafting procedures, limited quantity in some individuals and donor site morbidity have lead surgeons to look for alternative harvest sites or sources such as allograft or osteobiologics. Of these alternative harvest sites is the femoral shaft. Intramedullary contents from reaming are composed of bone marrow, and blood and bone spicules. In this respect, the reamed contents are similar to the bone routinely harvested from the iliac crest. Studies have shown that despite the reaming process using standard reamers, cells maintain their viability and are able to produce new bone. However, the addition of aspiration and irrigation used in the RIA system could potentially compromise the harvested cell viability and limit their osteogenic potential. In addition, Wenisch et al. have concluded that the harvested cells using standard intramedullary reamers not only proceed toward osteogenic differentiation, but also can be directed toward neurogenic differentiation. This suggests that reaming debris is a viable source of stem cells as well. RIA allows for these cells to be harvested. It is our hypothesis that the intramedullary contents harvested using the RIA system is similar to ICBG in cell viability and osteogenic potential.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 years or older
* Subjects undergoing a bone grafting procedure, either using an iliac crest or RIA system harvesting technique, or
* Subjects undergoing reamed femoral intramedullary nailing using the RIA reaming technique

Exclusion Criteria:

* Subjects under age 18
* Subjects with a history of: leukemia; cancer with bone metastases; renal failure, receiving dialysis; or on immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Project involves comparison of small samples taken from patients undergoing iliac crest or medullary reaming for comparison and review
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cell viability | 1 hour post-collection
Osteogenic potential | 1 hour post-collection

CONTACTS AND LOCATIONS:
Overall Officials: Brett D Crist, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No